CLINICAL TRIAL: NCT02690753
Title: A Turn and Positioning System and Standardized Incontinence Care Combined With Tailored Repositioning Versus a Standard Repositioning Protocol for Pressure Ulcer Prevention: A Multicenter Prospective Randomized Controlled Clinical Trial and Health Economical Analysis in a Hospital Setting
Brief Title: Pressure Ulcer Prevention: a Turn and Positioning System Combined With Incontinence Care and Tailored/Standard Repositioning
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Collaborators: Sage Products, LLC (Industry)
Responsible Party: Principal Investigator, UCVV, University Centre for Nursing and Midwifery, University Ghent
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PA2015/041
Record Dates: First submitted 2015-12-08; First posted 2016-02-24 (Estimated); Last update posted 2018-03-09 (Actual); Status verified 2018-03

CONDITIONS: Pressure Ulcers; Incontinence-associated Dermatitis
Keywords: Repositioning; Incontinence care; Prevention
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Tailored repositioning + Standardised incontinence care + TAP (Experimental): A protocol tailored to individual risk factors will be applied to patients at risk.Comfort Shield® barrier cream cloths will be used for incontinence care every morning and after each episode of incontinence. The Prevalon® Turn and Position System 2.0, SAGE will be used for turning and positioning patients at risk when laying in bed.
  Interventions: Procedure: A protocol tailored to individual risk factors; Device: The Prevalon® Turn and Position System 2.0; Device: Comfort Shield® barrier cream cloths
- Standard repositioning + Standardised incontinence care + TAP (Experimental): Instead of developing and using a tailored pressure ulcer prevention protocol, patients will receive standard care.Comfort Shield® barrier cream cloths will be used for incontinence care every morning and after each episode of incontinence. The Prevalon® Turn and Position System 2.0, SAGE will be used for turning and positioning patients at risk when laying in bed.
  Interventions: Device: The Prevalon® Turn and Position System 2.0; Device: Comfort Shield® barrier cream cloths
- Usual care (No Intervention): Instead of developing and using a tailored pressure ulcer prevention protocol, patients will receive standard care. Instead of using comfort Shield® barrier cream cloths, incontinence care will be given to patients using the standard procedure on the ward. Instead of using the turn and position system, patients will be turned according to the standard procedure on the ward.

INTERVENTIONS:
Procedure: A protocol tailored to individual risk factors
  Arms: Tailored repositioning + Standardised incontinence care + TAP
Device: The Prevalon® Turn and Position System 2.0
  Arms: Standard repositioning + Standardised incontinence care + TAP; Tailored repositioning + Standardised incontinence care + TAP
Device: Comfort Shield® barrier cream cloths
  Arms: Standard repositioning + Standardised incontinence care + TAP; Tailored repositioning + Standardised incontinence care + TAP

SUMMARY:
The prevalence of pressure ulcer in hospitals is 7,3% - 23%. The primary etiological factors are pressure or pressure combined with shear. Prevention is very important and comprises: preventive skin care including cleansing and protecting the skin from exposure to moisture, the systematic repositioning of the patient, the offloading of the heels from the surface of the bed, the use of adequate bed support surfaces and an adequate nutritional status. The development and implementation of a risk based prevention plan for individuals identified as being at risk is strongly recommended. Limited compliance exists towards pressure ulcer preventive interventions. 25,5% of the patients at risk receive fully adequate prevention in bed. The reposition frequence is adequate in 55% of patients at risk. There is a lack of rigorously performed research addressing the effectiveness of devices or risk based protocols to improve compliance. Health care budgets are limited, priorities should be set in the allocation of health care resources.

The primary aim of this study is to compare the effectiveness of the turn and position system (Prevalon®Turn and Position System 2.0, SAGE) versus standard care to improve reposition frequence in patients at risk. The second aim is to compare the effectiveness of a tailored protocol versus standard care to improve reposition frequence in patients at risk. The third aim is to compare the effectiveness of standardized incontinence care versus standard care to improve the incidence of pressure ulcers and incontinence-associated dermatitis (IAD). Also a health economic evaluation will be performed.

The study will be performed in hospital setting (university and general hospitals) in a random sample of 226 patients aged > 18 who are at risk of developing pressure ulcers. Patients will be recruited from three types of wards: intensive care units, geriatric wards and rehabilitation wards. Patients will be included in the study for a period of 8 days.

ELIGIBILITY:
Inclusion Criteria:

* At risk of developing pressure ulcers (Braden score < 17)
* Maximum 24hours admitted on the ward at the time of inclusion
* Expected lenght of stay: 8 days
* Free of pressure ulcers category II, II, IV and incontinence-associated dermatitis (IAD) category 2 at the start of the study

Exclusion Criteria:

- Patients with no active or supportive therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 227 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Turning compliance of nurses within the trial period as assessed by the researcher (unannounced) | within 8 days after the start of the study
  The researcher wil collect and administer data about turning compliance and compliance with the protocol

SECONDARY OUTCOMES:
Turning angle | within 8 days after the start of the study
  Per patient the researcher will measure two times the turning angle in which the patient is positioned.
Sacrum free of pressure | within 8 days after the start of the study
  Per patient the researcher will investigate two times if the sacrum is free of pressure while the patient is positioned.
Incidence of pressure ulcers and incontinence-associated dermatitis | within 8 days after the start of the study
Comfort and preferences of the caregiver | On baseline and at day 8 (the end of the study)
  Questions on comfort and preferences of the TAP, comfort shield barrier cream cloths and tailored repositioning will be assessed. At baseline these questions will assess the traditional care.
Comfort and tolerance of the patient | At day 8 (the end of the study)
  Questions on comfort and tolerance of the TAP, comfort shield barrier cream cloths and repositioning will be assessed by the caregiver. At baseline these questions will assess the traditional care.
Cost-effectiveness of the prevention of pressure ulcers | For the duration of the study (8 days)
  The following costs will be calculated to provide insight concerning cost-effectiveness:
  Objective time analysis of repositioning (by using a chronometer), Subjective time analysis of repositioning, Daily consumption of comfort shield barrier cream cloths and microclimate body pads

CONTACTS AND LOCATIONS:
Overall Officials: Dimitri Beeckman, PhD, Principal Investigator — University Ghent
Locations (15):
- Belgium (15):
  - AZ St. Maarten, Duffel, Antwerpen
  - AZ St. Dimpna, Geel, Antwerpen
  - AZ Nikolaas campus Beveren, Beveren, Oost-Vlaanderen
  - UZ Gent, Ghent, Oost-Vlaanderen
  - AZ Oudenaarde, Oudenaarde, Oost-Vlaanderen
  - ASZ Aalst, Aalst
  - AZ Monica, Antwerp
  - ZNA Hoge Beuken, Antwerp
  - ZNA St. Elisabeth, Antwerp
  - Imelda Ziekenhuis, Bonheiden
  - AZ St. Jan Brugge, Bruges
  - ASZ Geraardsbergen, Geraardsbergen
  - AZ Delta Menen, Menen
  - AZ St. Jan Oostende, Ostend
  - AZ Delta Roeselare, Roeselare

REFERENCES:
- [Background] Beeckman D, Van Damme N, Schoonhoven L, Van Lancker A, Kottner J, Beele H, Gray M, Woodward S, Fader M, Van den Bussche K, Van Hecke A, De Meyer D, Verhaeghe S. Interventions for preventing and treating incontinence-associated dermatitis in adults. Cochrane Database Syst Rev. 2016 Nov 10;11(11):CD011627. doi: 10.1002/14651858.CD011627.pub2. PMID 27841440
- [Background] Beeckman D, Van Lancker A, Van Hecke A, Verhaeghe S. A systematic review and meta-analysis of incontinence-associated dermatitis, incontinence, and moisture as risk factors for pressure ulcer development. Res Nurs Health. 2014 Jun;37(3):204-18. doi: 10.1002/nur.21593. Epub 2014 Apr 3. PMID 24700170
- [Derived] De Meyer D, Van Hecke A, Verhaeghe S, Beeckman D. PROTECT - Trial: A cluster RCT to study the effectiveness of a repositioning aid and tailored repositioning to increase repositioning compliance. J Adv Nurs. 2019 May;75(5):1085-1098. doi: 10.1111/jan.13932. Epub 2019 Jan 25. PMID 30549321
- See also: Website of the research group — http://www.ucvvgent.be